CLINICAL TRIAL: NCT04032860
Title: The Different Effects of Nucleotide and Nucleoside Analogues on the Prognosis of Hepatitis B Virus-Related Hepatocellular Carcinoma Patients After Curative Resection：a Randomized Controlled Trial
Brief Title: RCT of Different Effects of Nucleot(s)Ide Analogues on the Prognosis of HBV-HCC Patients After Curative Resection
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, linye he, doctor of liver surgery, Principal Investigator,, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1185022016
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: HCC; HBV Coinfection
Keywords: tenofovir, HBV, HCC, nucleo(t)side analogues, Entecavir
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ETV group (Experimental): group in which patients take ETV as antiviral therapy after curative treatment
  Interventions: Drug: Entecavir
- TDF group (Experimental): group in which patients take TDF as antiviral therapy after curative treatment
  Interventions: Drug: Tenofovir Disoproxil

INTERVENTIONS:
Drug: Tenofovir Disoproxil — patients with HBV-HCC would take TDF as antiviral therapy before curative treatment to see the prognosis after surgery
  Other Names: TDF
  Arms: TDF group
Drug: Entecavir — patients with HBV-HCC would take ETV as antiviral therapy before curative treatment to see the prognosis after surgery
  Other Names: ETV
  Arms: ETV group

SUMMARY:
In Asia, hepatocellular carcinoma (HCC) commonly occurred in the underlying hepatitis B virus (HBV)-related liver disease.Curative therapies could improve the prognosis of HCC patients. However, tumor recurrence after curative therapy remains high with a 5-year recurrence rate >70%.The risk for HCC development is increased for patient with HBV infection，but there was no consensus about which kind of oral antiviral treatment was the best option in the prevention of HBV related HCC recurrence after curative treatment.Therefore, we conducted this study to investigate the different effects of nucleotides(TDF) and nucleosides(ETV) on the prognosis of HBV-related HCC after curative resection.

DETAILED DESCRIPTION:
The study was designed to compare the efficacy of ETV and TDF for patients with HBV-related HCC patients undergoing curative liver resection. Eligible patients were randomly assigned in a 1:1 ratio via computer-generated allocation to either the ETV group or TDF group. A block size and strata were used in the randomization. In 2015, the American Association for the Study of Liver (AASLD) adopted ETV and TDF as first-line antiviral treatments for chronic hepatitis B. Patients in the ETV group received ETV tablets (RunZhong, CHIATAI TIANQING, China) 0.5 mg/d orally starting from 2-4 weeks before surgery; those in the TDF group receive TDF tablets(Viread, Aspen Port Elizabeth, China) 300 mg/d orally starting from 2-4 weeks before surgery. Antiviral treatment was continued unless there was unacceptable toxicity or withdrawal of consent.

Preoperatively, all patients underwent chest radiography and at least 2 dynamic imaging examinations (contrast-enhanced ultrasound, contrast-enhanced computed tomography(CT) or magnetic resonance imaging(MRI)). HBsAg and hepatitis B e antigen (HBeAg), HBV-DNA load, anti-HCV, alpha-fetoprotein (AFP), carcinoembryonic antigen(CEA), carbohydrate antigen 19-9(CA19-9), liver function and HBV genotypes were serologically examined within 1 week before surgery. Additional serum samples were collected to test single-nucleotide polymorphisms(SNPs) of the interleukin 28B(IL-28B) gene and serum levels of interferon(IFN)-λ1, IFN-λ2, IFN-λ3, IL-1β, tumor necrosis factor alpha(TNF-α), IL-6, IL-8 and IL-10. All serum and DNA samples were stored at -80°C until use.

After general anesthesia, surgery was performed as the standard protocol. Intraoperative ultrasonography was performed to assess the relationship of the tumor to vascular structures and to eliminate the extrahepatic metastasis. Pringle's maneuver was applied to occlude the blood inflow of the liver with cycles of 15 minutes clamp time and 5 minutes unclamped time. Liver resection was carried out by the Cusa Excel Ultrasonic Surgical Aspirator System(CUSA).

In the study, the primary outcome measures included both recurrence and overall survival rates from the date of the operation. Secondary outcome measures included patient tolerance of antiviral treatment, virologic response, liver function and additional cytokines such as IFN-λ1 IFN-λ2, IFN-λ3, IL-1β, TNF-α, IL-6, IL-8 and IL-10. All the patients received follow-up monitoring 1 month after the operation, every 3 months thereafter during the first 3 years, and then every 6 months in subsequent years. Physical examination, blood cell and differential counts, renal and liver function tests, AFP levels, HBV serology and HBV-DNA levels, serum IFN-λ level and imaging examinations were included in the follow-up examinations when necessary. Follow-up was continued until August 2020 when all surviving patients had a minimum follow-up of 24 months.

Tumor recurrence was diagnosed based on the identification of a new lesion on at least 2 radiological examinations and increased AFP levels (>100 ng/mL). Patients with tumor recurrence were actively treated with salvage liver transplantation, repeat hepatic resection, radiofrequency ablation, transcatheter arterial chemoembolization(TACE), sorafenib, and/or chemotherapy, depending on the extent of the disease, the liver function, and general condition of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years and less than 69 years old;
2. HBsAg positive HCV antibody negative and HIV antibody negative;
3. HBV-DNA>200 IU/mL;
4. BCLC（Barcelona Clinic Liver Cancer） staging O and A stage;
5. Platelet100×10^9/L;
6. Liver function Child-Pugh A,with no invasion in portal vein, hepatic vein and two large branches, no extrahepatic metastasis;
7. Creatinine clearance rate≥ 70 mL/min;
8. Antiviral treatment was not performed before surgery or antiviral treatment was accepted in a short term (<3 months);
9. No treatment was performed before the operation. The results of postoperatively histopathological biopsy were HCC;
10. The patients agree to participate in the clinical trial.

Exclusion Criteria:

1. The image found extrahepatic lymph nodes or visceral metastasis, the existence of large vascular invasion, the existence of bile duct embolus in the first operation;
2. The patient combined with a malignant tumor of other organs or had a history of other malignant tumors in other organs;
3. Liver function decompensation, such as: upper gastrointestinal bleeding, refractory ascites, coagulation dysfunction and so on;
4. contraindications to surgery;
5. Patients with poor compliance and not adhered to the follow-ups;
6. Patients refused to participate in the clinical trial.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1,3,5 years
  the difference of overall survival between two groups
Recurrence-free survival | 1,3,5 years
  the difference of overall survival between two groups

SECONDARY OUTCOMES:
cytokines | 1-3 years
  several cytokines secreted by patients after antiviral therapy such as interferon λ3
Viral reactivity | 1,3 year
  HBsAg，HBsAb，HBeAg，HBeAb，HBcAb

CONTACTS AND LOCATIONS:
Overall Officials: He Linye, Doctor, Principal Investigator — Westchina Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months of study completion
Access Criteria: requestors will be required to sign a data access agreement
URL: http://bethesda.org